CLINICAL TRIAL: NCT05543278
Title: Pragmatic Amiodarone Trial to Reduce Postoperative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Acronym: PATRONUS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Asishana A Osho, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022P001732
Record Dates: First submitted 2022-09-09; First posted 2022-09-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Surgery, Cardiac; Atrial Fibrillation
Keywords: Postoperative atrial fibrillation; POAF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amiodarone Arm (Experimental): In addition to the regular care provided to cardiac surgery patients, those in the Amiodarone Arm will also receive the amiodarone regimen.
  Interventions: Drug: Amiodarone
- Standard of Care Arm (No Intervention): Patients randomized to the Standard of Care Arm will receive the regular care provided to cardiac surgery patients.

INTERVENTIONS:
Drug: Amiodarone — Patients randomized to the Amiodarone Arm will receive a 5-day course of amiodarone after surgery.
  Arms: Amiodarone Arm

SUMMARY:
Postoperative atrial fibrillation is quite common after cardiac surgery with up to 1 in 3 patients experiencing this abnormal heart rhythm. Amiodarone, a medication commonly used to treat atrial fibrillation, has been previously shown to be an effective prophylactic agent at decreasing the occurrence of postoperative atrial fibrillation in patients who underwent coronary artery bypass surgery. However, despite many studies which have demonstrated its effectiveness, it has not been widely used due to the concern of side effects that can occur such as slow heart rate, low blood pressure, and lung toxicity. We have designed a study to test the effectiveness and safety of a short course of postoperative prophylactic amiodarone for patients undergoing non-coronary artery bypass cardiac surgery. We hypothesize that patients who receive the prophylactic amiodarone will have decreased rates of postoperative atrial fibrillation without significantly increased side effects compared to patients who receive the standard postoperative care after non-coronary artery bypass cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* All genders
* All non-coronary artery bypass cardiac surgery patients
* Preoperative normal sinus rhythm

Exclusion Criteria:

* Pre-existing atrial fibrillation or atrial arrhythmias
* Pre-existing heart block
* Cardiogenic shock
* Sick sinus syndrome
* Marked sinus bradycardia
* Preoperative amiodarone use
* Contraindication to amiodarone use

  * PR interval > 240 ms
  * QTc > 550 ms
  * 2nd or 3rd degree heart block
  * Liver impairment (INR > 1.7, AST/ALT > 2x normal)
  * Uncontrolled hyperthyroidism or hypothyroidism
  * Interstitial lung disease
  * Pregnancy and/or breastfeeding
  * Known hypersensitivity to any components of amiodarone, including iodine
* Emergent operation
* Planned MAZE or Pulmonary Vein Isolation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation | At least 1 minute duration, occurring before or on postoperative day 7
  The occurrence of postoperative atrial fibrillation detected by continuous telemetry, 12-lead electrocardiogram, and/or continuous ambulatory monitoring device through postoperative day 7.

SECONDARY OUTCOMES:
Operative mortality | Either in-hospital or within 30 days of procedure
  Operative mortality as defined by either in-hospital death or death within 30 days of discharge.
Stroke | Either in-hospital or within 30 days of procedure
  characterized by deficits lasting > 24 hours and/or imaging findings of infarction
Transient ischemic attack | Either in-hospital or within 30 days of procedure
  characterized by examination findings lasting < 24 hours without associated imaging findings
Electrical cardioversion | Either in-hospital or within 30 days of procedure
  Whether the patient required electrical cardioversion for hemodynamically unstable atrial fibrillation
Hemodynamic instability | Either in-hospital or within 30 days of procedure
  New hemodynamic instability (mean arterial pressure < 65 mmHg) after surgery
Initiation of systemic anticoagulation | Either in-hospital or within 30 days of procedure
  New indication of systemic anticoagulation for stroke prophylaxis due to atrial fibrillation
Myocardial infarction | Either in-hospital or within 30 days of procedure
  Myocardial infarction diagnosed based on ECG and laboratory testing including pursued intervention and/or findings from subsequent angiography will be compared between intervention groups. To be considered a myocardial infarction, the diagnosis will have to be confirmed and documented in the chart by a board-certified cardiologist.
Persistence of atrial fibrillation at discharge | Up to 90 days
  Atrial fibrillation as diagnosed by final ECG
Postoperative hospital length of stay | Up to 90 days
  The postoperative length of stay will be calculated starting from the end of the procedure to time of discharge.
Readmission | Within 30 days of procedure
  Rates of hospital readmission will be estimated for patients in each of the study intervention groups. Readmissions will be counted in this calculation if patients are admitted to the hospital. Emergency room visits without admission and outpatient visits will not count toward this calculation of readmission rates.
Symptomatic bradycardia | Either in-hospital or within 30 days of procedure
  Symptomatic bradycardia (HR < 55 bpm) requiring intervention
Number of patients with Amiodarone-related pulmonary toxicity | Either in-hospital or within 30 days of procedure
  Clinical diagnosis of amiodarone-related pulmonary toxicity that uses a combination of x-ray findings consistent with known amiodarone-related pulmonary toxicity and clinical findings including shortness of breath, non-productive cough, and other diagnoses have been excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Asishana A Osho, MD, MPH, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Greenberg JW, Lancaster TS, Schuessler RB, Melby SJ. Postoperative atrial fibrillation following cardiac surgery: a persistent complication. Eur J Cardiothorac Surg. 2017 Oct 1;52(4):665-672. doi: 10.1093/ejcts/ezx039. PMID 28369234
- [Background] Arsenault KA, Yusuf AM, Crystal E, Healey JS, Morillo CA, Nair GM, Whitlock RP. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003611. doi: 10.1002/14651858.CD003611.pub3. PMID 23440790
- [Background] Chatterjee S, Sardar P, Mukherjee D, Lichstein E, Aikat S. Timing and route of amiodarone for prevention of postoperative atrial fibrillation after cardiac surgery: a network regression meta-analysis. Pacing Clin Electrophysiol. 2013 Aug;36(8):1017-23. doi: 10.1111/pace.12140. Epub 2013 Apr 29. PMID 23627761
- [Background] Buckley MS, Nolan PE Jr, Slack MK, Tisdale JE, Hilleman DE, Copeland JG. Amiodarone prophylaxis for atrial fibrillation after cardiac surgery: meta-analysis of dose response and timing of initiation. Pharmacotherapy. 2007 Mar;27(3):360-8. doi: 10.1592/phco.27.3.360. PMID 17316148
- [Background] Lawton JS, Tamis-Holland JE, Bangalore S, Bates ER, Beckie TM, Bischoff JM, Bittl JA, Cohen MG, DiMaio JM, Don CW, Fremes SE, Gaudino MF, Goldberger ZD, Grant MC, Jaswal JB, Kurlansky PA, Mehran R, Metkus TS Jr, Nnacheta LC, Rao SV, Sellke FW, Sharma G, Yong CM, Zwischenberger BA. 2021 ACC/AHA/SCAI Guideline for Coronary Artery Revascularization: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 Jan 18;145(3):e18-e114. doi: 10.1161/CIR.0000000000001038. Epub 2021 Dec 9. No abstract available. PMID 34882435
- [Background] Colunga Biancatelli RM, Congedo V, Calvosa L, Ciacciarelli M, Polidoro A, Iuliano L. Adverse reactions of Amiodarone. J Geriatr Cardiol. 2019 Jul;16(7):552-566. doi: 10.11909/j.issn.1671-5411.2019.07.004. PMID 31447894
- [Background] Orr CF, Ahlskog JE. Frequency, characteristics, and risk factors for amiodarone neurotoxicity. Arch Neurol. 2009 Jul;66(7):865-9. doi: 10.1001/archneurol.2009.96. PMID 19597088
- [Background] Wolkove N, Baltzan M. Amiodarone pulmonary toxicity. Can Respir J. 2009 Mar-Apr;16(2):43-8. doi: 10.1155/2009/282540. PMID 19399307